CLINICAL TRIAL: NCT02668588
Title: A Multicentre, Double Blind, Randomized Placebo Controlled Trial to Assess the Effect of LF-PB on Seroma Formation in Women With Breast Cancer Undergoing Axillary Lymph Node Dissection
Brief Title: Extended-release of Octreotide (LF-PB) for the Treatment of Seroma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chemi S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LF-PB/14/05
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LF-PB 30 mg (Experimental): extended release of octreotide
  Interventions: Drug: extended release of octreotide
- Placebo (Placebo Comparator): extended release of placebo
  Interventions: Drug: extended release of placebo

INTERVENTIONS:
Drug: extended release of octreotide — 1 intramuscular injection of extended release of octreotide 30 mg
  Other Names: LF-PB 30 mg
  Arms: LF-PB 30 mg
Drug: extended release of placebo — 1 intramuscular injection of extended release of placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a multicentre, double blind, randomized placebo controlled trial to assess the effect of LF-PB on seroma formation in women with breast cancer undergoing Axillary Lymph Node Dissection (ALND).

Recruited patients will be randomly assigned to receive LF-PB 30 mg or placebo.

DETAILED DESCRIPTION:
The study will randomize between 24 and 72 subjects that received an ALND. A staged adaptive design is employed with two intermediate analyses and a final analysis. The first interim analysis at 24 treated subjects (at least 12 in each group) and the second at 48 treated subjects (at least 24 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Undergoing breast cancer surgery with axillary lymph node dissection during the current clinical trial;
* Negative serum pregnancy test for women of childbearing potential;
* Aspartate aminotransferase and alanine aminotransferase < 2 x the upper limit of normal;
* ECOG PS ≤ 1.

Exclusion Criteria:

* Previous axillary surgery on the same armpit (sentinel lymph node surgery is not exclusionary);
* Previous radiotherapy within five years from study drug administration on the same armpit undergoing surgery in this study;
* Concomitant participation to other clinical trial;
* Uncontrolled diabetes;
* Cholelithiasis;
* Human immunodeficiency virus or hepatitis B or C by screening serology;
* Uncontrolled hypothyroidism: if patient is being administered Eutirox/ Levothyroxine (or analogues) and levels of T3, T4 and TSH are confirmed to be within the normal ranges at screening, the patient can be enrolled in this study;
* Pregnant or lactating;
* Ascertained or presumptive hypersensitivity to the active principle and/or the ingredients of the study drug formulation;
* Corrected QT (using the Bazett formula, QTc) interval at screening or baseline > 450 msec (as the mean of 3 consecutive readings 5 minutes apart);
* Presence of any disease or use of concomitant medication known to increase the QT interval;
* Clinically significant or relevant abnormal medical history, vital sign, physical examination or laboratory evaluation finding;
* Corticosteroid treatment on a long-term basis (i.e. treatment for more than 3 consecutive days);
* Current or recurrent disease that could affect the results of the clinical or laboratory assessment required for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Incidence of seromas requiring an aspiration | Day 28 post surgery
  Subjects will undergo an echography at the operated axilla at every scheduled visit till Day 28 or until seroma resolution, whichever occurs first. In case of seroma presence the investigator will decide if an aspiration is required; the decision will be based on the clinical investigator's evaluation.
  In case of aspiration, the subject with seroma will be considered amenable for the statistical analysis of seroma incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Carcoforo, Prof., Principal Investigator — U.O. Clinica Chirurgica, A. O. Univ. Arcispedale S.Anna - Ferrara
Locations (7):
- Italy (7):
  - Az. Osp. Univ. Mater Domini, Catanzaro, Calabria
  - IRCCS Fondazione Pascale, Naples, Campania
  - Az. Osp. Univ. di Ferrara - Ospedale di Cona, Ferrara, Emilia-Romagna
  - Az.Osp. Univ. Policlinico di Modena, Modena, Emilia-Romagna
  - Az. Osp. Univ. di Parma, Parma, Emilia-Romagna
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genoa, Liguria
  - Az. Osp. Univ. Città Della Salute e Della Scienza di Torino, Turin, Piedmont

IPD SHARING:
Plan to Share IPD: Undecided